CLINICAL TRIAL: NCT06831695
Title: Comparison Between Surgical Outcomes of Craniotomy and Craniectomy Among Patients with Posterior Fossa Lesion
Brief Title: Comparison of Surgical Outcomes of Craniotomy and Craniectomy in Posterior Fossa Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Dr. Birat Thapa Magar, Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exp128
Record Dates: First submitted 2025-02-10; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Posterior Fossa Lesion
Keywords: Craniotomy; Craniectomy; Neurosurgery; Posterior Fossa; Brain Tumors
MeSH Terms: conditions — Brain Neoplasms | interventions — Craniotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Craniotomy (Active Comparator): This procedure involves creating a single free bone flap using high-speed drills. The bone is repositioned and secured using mini plates or sutures after the surgical intervention is completed. Post-operative monitoring will include assessment for CSF leakage, wound healing, and neurological recovery.
  Interventions: Procedure: Craniotomy
- Group B: Craniectomy (Active Comparator): In this approach, the bone is removed in pieces using rongeurs, leaving an open dural surface without replacement of the bone. The dura is closed with sutures, and dural augmentation may be performed as needed. Post-operative assessment will focus on complications such as pseudomeningocele, CSF leakage, and extended hospital stays.
  Interventions: Procedure: Craniectomy

INTERVENTIONS:
Procedure: Craniotomy — Intervention: Bone flap replaced after dural closure Additional Information: This procedure involves creating a single free bone flap using high-speed drills. The bone is repositioned and secured using mini plates or sutures after the surgical intervention is completed. Post-operative monitoring will include assessment for CSF leakage, wound healing, and neurological recovery.
  Arms: Group A: Craniotomy
Procedure: Craniectomy — Intervention: Bone permanently removed Additional Information: In this approach, the bone is removed in pieces using rongeurs, leaving an open dural surface without replacement of the bone. The dura is closed with sutures, and dural augmentation may be performed as needed. Post-operative assessment will focus on complications such as pseudomeningocele, CSF leakage, and extended hospital stays.
  Arms: Group B: Craniectomy

SUMMARY:
The purpose of this randomized controlled trial is to compare the surgical outcomes of craniotomy and craniectomy among patients with posterior fossa lesions. The study aims to determine differences in post-operative complications, hospital stay duration, and patient recovery between the two surgical techniques.

DETAILED DESCRIPTION:
Patients diagnosed with posterior fossa lesions will be randomly assigned into two groups. Group A will undergo craniotomy, where the bone flap is replaced after dural closure, while Group B will undergo craniectomy, where the bone is permanently removed. Outcomes will be assessed based on post-operative complications such as CSF leakage, pseudomeningocele formation, post-operative headache, and length of hospital stay. The study aims to provide evidence to determine the superior surgical approach in terms of patient outcomes and healthcare cost reduction.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with posterior fossa lesions
* Age range: 7-70 years
* Patients with cerebellar hematoma (traumatic or spontaneous)

Exclusion Criteria:

* Previous posterior fossa surgery
* Brainstem hematoma
* Tumors involving the overlying dura or bone

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-04 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of CSF leakage | Up to 6 months post-surgery
  Definition: CSF leakage is defined as the presence of clear fluid discharge from the surgical site, confirmed via clinical examination and biochemical analysis of β-2 transferrin.
  Measurement: Evaluated by clinical assessment at routine follow-ups and imaging studies when indicated.
Occurrence of pseudomeningocele | Up to 6 months post-surgery
  Definition: Pseudomeningocele is defined as an abnormal collection of cerebrospinal fluid in the surgical site, detected through physical examination and confirmed by imaging techniques such as MRI or CT scan.
  Measurement: Follow-up visits at 1, 3, and 6 months post-surgery.
Severity of post-operative headache | Immediately post-surgery, at 3 months, and at 6 months post-surgery
  Definition: Post-operative headache will be assessed using the Catalano grading system, categorizing severity from 0 (no headache) to 4 (severe, refractory to medication).
  Measurement: Self-reported patient evaluations at each follow-up visit.
Length of hospital stay | From immediate post-surgery until hospital discharge, assessed up to 4 weeks
  Definition: The total number of days a patient remains hospitalized post-surgery, including any extended stay due to complications.
  Measurement: Recorded from hospital admission to discharge.

IPD SHARING:
Plan to Share IPD: Undecided